CLINICAL TRIAL: NCT02184481
Title: Working Memory Training to Decrease Depression, Anxiety and Rumination in Dysphoric Students
Brief Title: Working Memory Training for Dysphoric Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Ingmar Franken, Professor, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Franken 5
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Depression
Keywords: Depression; Anxiety; Working memory; Rumination; Cognitive training; Executive functioning
MeSH Terms: conditions — Depression; Anxiety Disorders; Rumination Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Working memory training (Experimental): Participants executed the training for three weeks, three times a week, half an hour per session. The training was a game in which the participant was a person who had to become strong to fight with a fantasy figure. The person could become stronger when giving the right answers in eight different working memory tasks. The level adapted to the working memory capacity of the participant.
  Interventions: Behavioral: Working memory training
- Placebo training (Placebo Comparator): Participants executed the training for three weeks, three times a week, half an hour per session. The training was a game in which the participant was a person who had to become strong to fight with a fantasy figure. The person could become stronger when giving the right answers in eight different working memory tasks. The level in the placebo condition was easy and did not adapt to the working memory capacity of the participant.
  Interventions: Behavioral: Placebo training

INTERVENTIONS:
Behavioral: Working memory training
  Arms: Working memory training
Behavioral: Placebo training
  Arms: Placebo training

SUMMARY:
Depression is associated with impairments in executive functions, including working memory (WM) which is needed to maintain and manipulate goal-relevant information. Due to these WM impairments depressed individuals have difficulties inhibiting and shifting from irrelevant (negative) information and updating goal relevant information. This study explored whether training WM decreases these impairments and reduces clinical symptoms of depression, anxiety and rumination. Sixty-one students with an elevated score on the BDI-II, representing a dysphoric mood state, executed a working memory training (n = 34) or placebo training (n = 27). Before and after training their depression, anxiety, rumination and working memory were assessed. Furthermore, they executed a working memory task while their pupil dilation was measured to assess their fatigue. Moreover, the investigators compared the dysphoric students with a healthy student population on all measures.

ELIGIBILITY:
Inclusion Criteria:

* BDI 10 of higher for dysphoric group
* BDI 5 or lower for healthy control group

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2013-09; Primary Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory Second Edition (BDI-II) score change between pre and post measurement | Pre training (baseline), post training (4 weeks after baseline, training starts 1 day after baseline)
  Depression is measured with the BDI-II

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) scores change from pre to post training measurement | Pre training (baseline), post training (4 weeks after baseline, training starts 1 day after baseline)
  The STAI measures state, trait and total anxiety

OTHER OUTCOMES:
Ruminative Response Scale (RRS) score change between pre and post training | Pre training (baseline), post training (4 weeks after baseline, training starts 1 day after baseline)
  The RRS measures rumination
Spanboard task | Pre training (baseline), post training (4 weeks after baseline, training starts 1 day after baseline)
  The Spanboard task measures working memory capacity
N-back task | Pre training (baseline), post training (6 weeks after baseline, training starts 1 day after baseline)
  The n-back task was assessed while participants pupil dilation was measured with the eyetracker. The aim of this measurement was to measure fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus University Rotterdam, Rotterdam, South Holland, Netherlands

REFERENCES:
- [Derived] Hopstaken JF, Wanmaker S, van der Linden D, Bakker AB. Does Dysphoria Lead to Divergent Mental Fatigue Effects on a Cognitive Task? PLoS One. 2015 Jun 15;10(6):e0130304. doi: 10.1371/journal.pone.0130304. eCollection 2015. PMID 26075389